CLINICAL TRIAL: NCT06580262
Title: Evaluation of the Vittel Criteria for Pre-hospital Triage of Severe Trauma Patients in the French West Indies and in French Guiana
Acronym: TRAUMA-DOM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 22_RIPH3-12
Record Dates: First submitted 2024-08-22; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Severe Trauma
Keywords: Trauma; Severe trauma; Vittel criteria; Hospital emergency; Triage score
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of severe trauma treated in the emergency departments: Patients suspected of severe trauma defined as trauma likely to have caused multiple injuries and/or threatening the vital or functional prognosis.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — The investigator takes care of the patient according to the protocol in force in his department and decides on the final orientation of the patient (transfer to intensive care unit/ICU, hospitalization or home discharge).
  No recommendations or instructions are given to the investigators. Each investigator is free to decide on his care and the terms of transfer, hospitalization and discharge.

SUMMARY:
Severe trauma is a public health problem because it is the leading cause of death in young people and the third leading cause of death in France for all ages. These injuries will cause anatomical and functional after-effects that are sometimes permanent, and are therefore among the leading causes of acquired disability in France.

The Vittel criteria constitute a decision-making algorithm of 24 criteria for triage of trauma patients. The presence of only one criterion out of the 24 must direct the patient to a trauma referral center. The existence of only one trauma referral center per territory questions the relevance of using the Vittel criteria in the French Antilles and Guiana.

It therefore seems important that the relevance of the different Vittel criteria be reassessed in our territories, where the typology of patients and the urban network is different compared to that of mainland France. are a common cause of severe trauma, followed by assaults or fights, accidents at work, during leisure or at home, falls from a great height, and weapon-related injuries. Special and rapid care is then necessary.

This is why trauma severity criteria and triage scores are used to target these serious patients and direct them to the appropriate healthcare facilities.

The Vittel criteria constitute a decision-making algorithm of 24 criteria for triage of trauma patients. The presence of only one criterion out of the 24 must direct the patient to a trauma referral center. The existence of only one trauma referral center per territory questions the relevance of using the Vittel criteria in the French Antilles and Guiana.

It therefore seems important that the relevance of the different Vittel criteria be reassessed in Martinique, Guadeloupe and french Guiana, french overseas territories, where the typology of patients and the urban network is different compared to that of mainland France.

DETAILED DESCRIPTION:
Trauma severity criteria and prehospital triage scores have been proposed since the 1990s. In 2002, a conference of experts in France proposed a decision algorithm for prehospital triage of trauma patients, known as the Vittel criteria. Indeed, the presence of a single criterion out of the 24 others should direct the patient to a trauma referral center (Level 1 Trauma Center). However, since their implementation, few studies have evaluated the relevance of these criteria on over- or under-triage, on the prescription of additional imaging tests, and finally on the prognosis of patients, including disabling sequelae. Indeed, some criteria are subjective and taken alone, it seems difficult to be able to put them on the same level to guide the patient.

In the French Antilles-Guiana inter-region, trauma from accidents on public roads and assaults with knives or firearms are a very common reason for interventions by SMUR teams. Despite this frequency, knowledge of the local epidemiology of these injuries is patchy. Furthermore, the referral of patients treated in pre-hospital care, either by firefighter teams or by the SMUR, is almost always done to the only reference health facility in each of the three French departments (Martinique, Guadeloupe, Guiana). The existence of only one trauma reference center per territory questions the relevance of using the Vittel criteria in the French Antilles-Guyana.

Twenty years after the development of the Vittel criteria, several changes have occurred in society, particularly in road safety and personal protective equipment. These advances would result in a reduction in the risks and severity related to accidents. Despite all these security advances, there is a lack of use and respect for them in the territories of the Antilles-Guiana. At the same time, violence and assaults by weapon have evolved with the use of firearms and weapons of war relatively frequently in our territories.

The relevance of the various Vittel criteria must be reassessed, particularly in the Antilles-Guyana where the typology of patients and the urban network is different from that of mainland France. The hypotheses are that certain criteria such as age, comorbidities, speed and deformation of vehicles, taken in isolation, would not be prognostic criteria for a serious anatomical injury or intensive care or even early mortality. Conversely, other criteria such as the taking of toxics or two-wheeled road accidents would be more important criteria to take into consideration.

ELIGIBILITY:
Inclusion Criteria:

* Minor patients (2-17 years) and adults (≥ 18 years).
* Patients treated in the emergency units of the hospitals participating in the study, whether they were brought by a SAMU/SMUR team, by a rescue and victim assistance vehicle or arrived directly.
* Patients suspected of severe trauma, defined as trauma likely to have caused multiple injuries and/or threatening the vital or functional prognosis.
* Patient if he is able to, or representative of the patient in case of incapacity, having given his agreement for the use of his medical data for this research.

Exclusion Criteria:

* Absence of consent from the patient, or representative to the use of the data for the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of severe trauma, treated in the emergency units of the hospitals participating in the study (Martinique, Guadeloupe, Frech Guiana).
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To compare the frequency of each Vittel criterion according to the patient's status within 30 days | 30 days
  Calculation of the proportion of each Vittel criterion in the two groups defined according to the patient's status at day 30 (alive vs. deceased or hospitalized in intensive care).

SECONDARY OUTCOMES:
To compare the discriminatory capacity of the different Vittel criteria to estimate the probability of occurrence of a serious anatomical lesion in severely traumatized patients treated by the SAMU/SMUR of the French Antilles-Guiana | 13 months
  Calculation of the area under the ROC curve of the different Vittel criteria to evaluate a posteriori their performance in predicting, in severely traumatized patients, a serious anatomical lesion defined by an ISS score > 15.
To compare the discriminatory capacity of the different Vittel criteria to estimate the probability of having to resort to a massive transfusion in severely traumatized patients treated by the SAMU/SMUR of the French Antilles-Guiana | 13 months
  Calculation of the area under the ROC curve of the different Vittel criteria to evaluate a posteriori their performance in predicting a massive transfusion (defined by 5 red blood cell concentrates (RBCs) in 3 hours or 8 RBCs in 6 hours or 10 RBCs in 24 hours).
To assess the feasibility of having firefighters fill out a form to collect among the Vittel criteria those relating to the physical circumstances of the accident | 13 months
  Proportion of files for which the "physical circumstances of the accident" sheet was completed by the firefighters.

CONTACTS AND LOCATIONS:
Overall Officials: Papa Gueye, PhD, Principal Investigator — University Hospital Center of Martinique
Locations (2):
- France (2):
  - Hospital of Cayenne, Cayenne, French Guiana
  - University Hospital Center of Guadeloupe, Pointe à Pitre, Guadeloupe